CLINICAL TRIAL: NCT07013682
Title: Platelet Rich Fibrin Adjunctive to Non-surgical Periodontal Therapy: a 6-month Split-mouth Randomized Controlled Clinical Trial
Brief Title: PRF as Adjunct to Subgingival Instrumentation in Step 2 Periodontal Therapy
Acronym: PRFSTEP2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRF2
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Periodontitis; Periodontal Inflammation; Periodontal Attachment Loss
MeSH Terms: conditions — Periodontitis; Periodontal Attachment Loss | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: This is a split-mouth study. One side of the mouth (upper and lower jaw) will be treated with adjunctive PRF during non-surgical mechanical therapy and the other without.
Who Masked: Participant, Outcomes Assessor
Masking Description: Opaque sealed envelopes will held the randomisation key of which side has to be treated with PRF. After completion of the non-surgical mechanical debridement in the whole dentition, the sealed envelope will be opened. PRF will be obtained from the elbow vene and after centrifugation the PRF will be applied in the pockets ≥ 5 mm. On the control side an empty cannula will be held.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control side (Sham Comparator): After non-surgical mechanical debridement of all pockets ≥ 5 mm, an empty syringe will be inserted.
  Interventions: Biological: Control, non-surgical mechanical debridement alone
- Test side (Active Comparator): After non-surgical mechanical debridement of all pockets ≥ 5 mm, PRF will be inserted.
  Interventions: Biological: PRF as adjunct to non-surgical mechanical debridement

INTERVENTIONS:
Biological: PRF as adjunct to non-surgical mechanical debridement — Non-surgical mechanical debridement with hand and power-driven instruments will be performed. Venous blood will be harvested from the patient and centrifuged. Immediately afterwards, the PRF will be inserted in all pockets of the allocated side of the jaw in all pockets ≥ 5 mm.
  Arms: Test side
Biological: Control, non-surgical mechanical debridement alone — Non-surgical mechanical debridement with hand and power-driven instruments will be performed. Venous blood will be harvested from the patient and centrifuged. Immediately afterwards, an empty sy will be inserted in all pockets of the allocated control side of the jaw in all pockets ≥ 5 mm.
  Arms: Control side

SUMMARY:
Periodontitis is characterized by a chronic, multifactorial inflammatory process driven by dysbiotic plaque biofilms. It is recognized as the most common chronic inflammatory non-communicable disease in humans. The advanced and severe forms of periodontitis have an estimated prevalence of 7.4%, while milder forms can affect up to 50% of the population.

If left untreated, periodontitis can lead to tooth loss. However, it is largely preventable and treatable with mechanical non-surgical periodontal therapy. To improve periodontal healing and thus clinical attachment gain after non-surgical therapy, adjunctive bioactive formulations such as enamel matrix derivatives, sodium hypochlorite, locally delivered antimicrobials, or hyaluronic acid have recently been proposed. However, these agents are non-autologous formulations and expensive.

Platelet-rich fibrin (PRF) acts as a scaffold that inhibits the early migration of epithelial cells into the periodontal tissues. Its regenerative properties are primarily due to its ability to promote angiogenesis. This ability is attributed to the 3D fibrin matrix, which can simultaneously transport several cytokines and growth factors. These include vascular endothelial growth factor (VEGF), insulin growth factor (IGF), transforming growth factor β1 (TGF-β1) and platelet-derived growth factor (PDGF). PRF further shows antibacterial properties and accelerates soft tissue healing. So far PRF is not routinely used in periodontal non-surgical therapy.

The aim of this 6-month, split-mouth randomized clinical trial including 20 patients is to test whether PRF can improve the results after non-surgical therapy.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether scaling and root planing (SRP) combined with the application of a platelet-rich fibrin (PRF) membrane can improve clinical outcomes. Specific outcomes to be measured include reduction in probing pocket depth (PPD), gain in clinical attachment level (CAL), improvement in plaque index, gingival index, and minimization of gingival recession (GR) compared to SRP therapy alone after 3 and 6 months. Further patients reported pain outcomes as well as bacterial profiles and inflammatory markers will be checked.

Patients presenting with periodontitis stage II-IV will be included having at least 20 teeth.

The study includes multiple timepoints: a screening visit, a visit for full-mouth non-surgical treatment with and without PRF in a split-mouth design, a 7-day follow-up visit, a 3-month follow-up visit, and a final assessment 6 months after the non-surgical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years
* Periodontitis stage II-IV, grade A/B/C, generalized
* Presence of at least 20 teeth (excluding wisdom teeth)
* Absence of removable dentures
* Patients willing to provide written informed consent and to complete the 6- month study follow-up

Exclusion Criteria:

* Patients already participating in other clinical trials
* Periodontal treatment in the previous 12 months
* Antibiotic treatment 3 months prior to study entry
* Antibiotic prophylaxis required for dental treatment
* Current use of any medication that may affect the clinical features of periodontitis
* Pregnant/lactating
* Any condition that prevents venipuncture
* Not willing to venous puncture
* Current cancer treatment
* History of radiation in the head-neck area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Change in PPD after 6 months | 6 months follow-up
  Changes in probing depths measured with a periodontal probe in mm from baseline to 6 months after non-surgical periodontal therapy

SECONDARY OUTCOMES:
Change in PPD after 3 months | 3 months follow-up
  Changes in probing depths measured with a periodontal probe in mm from baseline to 3 months after non-surgical periodontal therapy
Change in clinical attachment level (CAL) | 3 months and 6 months follow-up
  The distance in millimeters from the cement-enamel junction (CEJ) to the bottom of the periodontal pocket. This will be assessed using a periodontal probe with mm scale
Frequency of residual pockets | 3 months and 6 months follow-up
  The number of probing depth of > 5 mm will be assessed
Full-mouth bleeding score (FMBS) | Baseline, 3 months and 6 months follow-up
  Percentage of tooth sites (six sites) revealing the presence of bleeding on probing to the bottom of the periodontal pocket. For this a periodontal probe with mm scale will be used, a score of 0% will represent perfect hygiene and 100% plaque on all surfaces (worst value)
Gingival Recession (REC) | Baseline, 3 months and 6 months follow-up
  The distance in millimeters from the gingival margin to the cemento-enamel junction (CEJ). The measurements will be performed with a periodontal probe with a mm scale
Comparison in PPD change between smokers and non-smokers | 3 months and 6 months follow-up
  Differences in outcome measures will be assessed
Levels of periodontal bacteria | Baseline, 3 months and 6 months follow-up
  Levels of periodontal bacteria will assessed by multiplex Polymerase Chain Reaction
Comparison of periodontal bacteria between smokers and non-smokers | Baseline, 3 months and 6 months follow-up
  Levels of periodontal bacteria will assessed by multiplex PCR
Levels of Interleukin (IL)-1beta | Baseline, 7 days, 3 months and 6 months follow-up
  Levels in gingival crevicular fluid will be assessed with ELISA assays
Levels of Matrix metalloproteinase (MMP)-8 | Baseline, 7 days, 3 months and 6 months follow-up
  Levels in gingival crevicular fluid will be assessed with ELISA assays
Levels of IL-8 | Baseline, 7 days, 3 months and 6 months follow-up
  Levels in gingival crevicular fluid will be assessed with ELISA assays
Comparison between smokers and non-smokers in levels of IL-1beta | Baseline, 7 days, 3 months and 6 months follow-up
  Levels in gingival crevicular fluid will be assessed with ELISA assays
Comparison between smokers and non-smokers in levels of MMP-8 | Baseline, 7 days, 3 months and 6 months follow-up
  Levels in gingival crevicular fluid will be assessed with ELISA assays
Comparison between smokers and non-smokers in levels of IL-8 | Baseline, 7 days, 3 months and 6 months follow-up
  Levels in gingival crevicular fluid will be assessed with ELISA assays
Antimicrobial activity of PRF | At visit of Step-2 therapy, expected to be ca. 2-4 weeks after baseline
  Remnants of PRF will be used for assessment of antimicrobial activity
Comparison between smokers and non-smokers in antimicrobial activity of PRF | At visit of Step-2 therapy, expected to be ca. 2-4 weeks after baseline
  Remnants of PRF will be used for assessment of antimicrobial activity
Patient reported pain outcomes | Each day from day 1 to 7 after non-surgical periodontal therapy
  A visual analogue scale (100 mm) will be used for the left and right side of the jaw to quantify pain levels. 0 will be no pain at all and 100 mm the worst imaginable level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Salvi, DMD, Principal Investigator — University of Bern
Locations (1):
- Department of Periodontology, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No